CLINICAL TRIAL: NCT04899102
Title: Pilot Study of Time-Restricted, Intermittent Fasting for Non-Alcoholic Fatty Liver Disease in Non-Obese Adults
Brief Title: Intermittent Fasting for NAFLD in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kathleen E Corey, Director, Fatty Liver Clinic Assistant Professor, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P002672
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Fatty Liver; Intermittent Fasting; Fatty Liver, Nonalcoholic; Non-Alcoholic Fatty Liver Disease; Liver Fat
Keywords: Fatty Liver; Intermittent Fasting; Non-obese; Diet; Nutrition; Time-restricted; Liver Fat; Non-Alcoholic Fatty Liver Disease; Fatty Liver, Nonalcoholic
MeSH Terms: conditions — Fatty Liver; Intermittent Fasting; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Every individual enrolled will follow a special type of diet for 6 weeks, called time-restricted, intermittent fasting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Time-Restricted, Intermittent Fasting Group (Experimental): Special type of diet for 6 weeks, called time-restricted, intermittent fasting.
  Interventions: Behavioral: Time-Restricted, Intermittent Fasting

INTERVENTIONS:
Behavioral: Time-Restricted, Intermittent Fasting — A special type of diet for 6 weeks, called time-restricted, intermittent fasting.

SUMMARY:
NAFLD is a growing threat to public health. Currently, there is a significant need for highly effective treatments for NAFLD. Non-obese NAFLD (BMI<30kg/m2) is an increasingly recognized condition, sometimes described as "lean NAFLD". Intermittent Fasting (IF) may be uniquely beneficial in non-obese NAFLD. The purpose of this study is to identify non-pharmacologic, lifestyle-based methods of NAFLD treatment within non-obese adults.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD), which encompasses a spectrum from simple steatosis and steatohepatitis (NASH) to fibrosis and cirrhosis, is the leading cause of liver disease in the United States. There are currently no FDA-approved pharmacologic therapies for NAFLD and NASH, and standard low-calorie diets are often minimally effective, difficult to adhere to and to maintain. Thus, continued investigation of strategies to treat NAFLD and NASH is greatly needed. Non-obese NAFLD (BMI<30kg/m2) is an increasingly recognized condition, sometimes described as "lean NAFLD". It is estimated that 10-20% of American and Europeans without obesity have this condition. There is a pressing need for the study of lifestyle interventions independent of weight loss to treat this important subset of NAFLD patients. This protocol aims to investigate the utility of time restricted, intermittent fasting (TRF) as a potential method. Adults with non-obese NAFLD are at risk of progression to end-stage liver disease and development of cardiometabolic disease. Intermittent Fasting (IF) may be uniquely beneficial in non-obese NAFLD. IF is characterized by periods of dietary restriction leading to metabolic production and use of ketones from adipocytes rather than hepatically-derived glucose.

The goal of this study is to learn if time-restricted, intermittent fasting can help reduce the amount of fat in the liver in adults with non-alcoholic fatty liver disease (NAFLD). Ideally, this study will yield more information about time-restricted, intermittent fasting as a potential lifestyle-based treatment for adults with NAFLD and a body mass index (BMI) between 23-30 kg/m^2.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Age 18 years or older at time of consent
3. BMI 23-30kg/m^2 at screening
4. Evidence of NAFLD confirmed by historical procedure obtained no more than 6 months prior to the screening visit, defined as:

   * Grade >=1 steatosis on clinical liver biopsy; OR
   * Fatty liver on validated imaging modality (non-contrast CT scan, MR Spectroscopy, MRI proton density fat fraction, ultrasound)
5. Liver fat fraction ≥10% on H-MRS performed during the screening period
6. Hepatitis C antibody and Hepatitis B surface antigen negative at screening

Exclusion Criteria:

1. Heavy alcohol use for at least 3 consecutive months within the past 5 years prior to screening [heavy alcohol consumption is defined as: > 20g daily for women or > 30mg daily for men, assessed by the Lifetime Drinking History assessment at screening (23, 24)].
2. Evidence of other known forms of chronic liver disease including:

   • Alcoholic liver disease, hepatitis B, hepatitis C, PBC, PSC, autoimmune hepatitis, Wilson disease, iron overload, alpha-1-antitrypsin deficiency, drug-induced liver injury, known or suspected hepatocellular carcinoma (HCC).
3. Current or prior history of Type II Diabetes requiring insulin or sulfonylureas due to risk of hypoglycemia with fasting.
4. Use of any pharmacological treatments for NAFLD/NASH within the 6 months prior to the screening visit, except vitamin E. Patients on a stable dose of vitamin E can be enrolled in the study.
5. Unstable body weight [defined as: >10% reduction in body weight in the 6 months prior to the screening visit]
6. Known cirrhosis, stage 4 fibrosis on prior liver biopsy, or clinical evidence of cirrhosis or portal hypertension on imaging or exam.
7. Current or prior history of Child-Pugh score ≥7.
8. History of liver transplant, or current placement on a liver transplant list.
9. Known positivity for human immunodeficiency virus infection.
10. Prior or planned bariatric surgery, patients on active pharmacological treatment for weight loss, or active involvement in a weight loss program.
11. Routine MRI exclusion criteria, such as the presence of a pacemaker or cerebral aneurysm clip.
12. Chronic Kidney Disease (CKD) with eGFR < 60.
13. For women of child-bearing potential (WOCBP): positive urine hCG, trying to achieve pregnancy, or breastfeeding [a negative urine pregnancy test is required at screening for women of child-bearing potential].
14. Other medical conditions or severe chronic illnesses that, in the opinion of the Investigator, may present a contraindication to study participation.
15. Any other condition that, in the opinion of the Investigator, may hinder study compliance or completion of the study schedule of assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Liver Fat Content | change from baseline to 6 weeks
  Liver Fat Content as measured by hydrogen-magnetic resonance spectroscopy (H-MRS)

SECONDARY OUTCOMES:
≥30% Relative Liver Fat Reduction Proportion | change from baseline to 6 weeks
  Proportion of subjects with a ≥30% relative reduction in hepatic fat
Visceral Adipose Tissue Content | change from baseline to 6 weeks
  Visceral Adipose Tissue Content as measured by magnetic resonance imaging/magnetic resonance spectroscopy (MRI/MRS)
Quality of Life Score | change from baseline to 6 weeks
  Quality of Life Score as measured by Chronic Liver Disease-NAFLD questionnaire (CLDQ-NAFLD)
Dietary Intake | change from baseline to 6 weeks
  Dietary Intake as measured by caloric intake and nutrient contents, assessed by ASA24

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Corey, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Final Research Data, with all patient identifiers removed, will be available to other researchers through request to the PI. Because information contained in the final research data will include multiple demographic and biological variables that could potentially be used in concert to identify participants, it will be shared only under a Data Sharing Agreement that includes (1) a commitment to using the data only for research purposes and not to identify any individual participant and (2) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol